CLINICAL TRIAL: NCT04034797
Title: AmbulaNCE Teletransmited PHOtography for Trauma REgulation
Acronym: NiCEPHORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2019-A00137-50
Record Dates: First submitted 2019-03-27; First posted 2019-07-26 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2020-09

CONDITIONS: Trauma; Telemedicine
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photo (Experimental)
  Interventions: Other: Photography teletransmission
- No photo (Active Comparator)
  Interventions: Other: No photo

INTERVENTIONS:
Other: Photography teletransmission — A photography of the trauma is teletransmitted to SAMU's physician
  Arms: Photo
Other: No photo — Usual management without photography teletransmission
  Arms: No photo

SUMMARY:
Physicians in charge of medical regulation within French SAMU have to take difficult decisions regarding patient's orientation (in or out-of hospital care) but suffer from lack of information. Such information usually consist in a simple phone conversation without any visual information. Visual assesment of the situation would be of great help, especially for traumatized patients.

Private Ambulance societies all over territory in charge of SAMU 86 now work with teletransmission devices allowing photography transmission.

The objective of the study is to determine if routine use of teletransmitted photography help SAMU 86's physians for a better orientation of non-severe traumatized patients, especially by avoiding unnecessary transportations to Emergency Departments.

ELIGIBILITY:
Inclusion Criteria:

* Emergency call at SAMU for trauma issue
* Pre-hospital management by private ambulance equipped with teletransmission device

Exclusion Criteria:

* Severe trauma with need of a pre-hospital emergency medical team
* Traffic accident
* Head trauma associated with anticoagulant therapy or platelet antiagregant therapy
* Pre-hospital management by firefighters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Impact of Photography on patient orientation | 1 - 2 hours
  Number of patient dispatched anywhere else than the local hospital after ambulance assesement.
  Either the patient was dispatched to a higher level hospital (i.e. if the local hospital doesn't provide surgical facility when the patient needs it) or he was leaved at home and oriented to a general practitioner.

SECONDARY OUTCOMES:
Undertriage | 10 days
  To evaluate the number of patients initially oriented to out-of hospital care that needed to go to emergency department during following days
Overtriage | 10 days
  To evaluate the number of patients initially oriented to in-hospital care when it wasn't necessary

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magimel-Pelonnier E, Marjanovic N, Couvreur R, Drugeon B, Mimoz O, Guenezan J. Photography tele-transmission by regular ambulance staff for the management of mild traumatic injury: the NiCEPHORE randomised-controlled trial. Scand J Trauma Resusc Emerg Med. 2022 Oct 14;30(1):53. doi: 10.1186/s13049-022-01026-0. PMID 36242052